CLINICAL TRIAL: NCT05411861
Title: Randomized, Double-Blind, Placebo- and Active-Controlled, Dose Escalation and Optional Dose Expansion Study to Evaluate Safety, Efficacy, and PK of CPL-01 in Post-Op Pain After Unilateral Distal First Metatarsal Bunionectomy + Osteotomy
Brief Title: Post-Operative Pain and Opioid Reduction Trial After Bunionectomy
Acronym: MERIT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cali Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CPL-01-202
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Hallux Valgus and Bunion
MeSH Terms: conditions — Hallux Valgus; Bunion | interventions — Analgesics, Non-Narcotic

STUDY DESIGN:
Intervention Model Description: Bunion Surgery
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Separate blinded and unblinded study teams
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CPL-01 (Experimental): Low dose of CPL-01
  Interventions: Drug: Analgesic Non Narcotic
- Ropivacaine HCl (Active Comparator): Low dose of Ropivacaine HCl
  Interventions: Drug: Analgesic Non Narcotic
- Placebo (Placebo Comparator): Low volume of placebo
  Interventions: Drug: Analgesic Non Narcotic

INTERVENTIONS:
Drug: Analgesic Non Narcotic — Injection of protocol-specified volume of local analgesic
  Other Names: Infiltration of local analgesic

SUMMARY:
This is a Phase 2b, randomized, double blind, placebo and active controlled study with an Ascending Dose Stage and an optional Dose Expansion Stage in subjects undergoing bunionectomy.

DETAILED DESCRIPTION:
Near the completion of surgery, a single dose of study drug (CPL-01, saline placebo, or ropivacaine HCl) will be infiltrated. Subjects will remain in the hospital/research facility for a minimum of 72 hours after the start of study drug administration to undergo postoperative assessments. Subjects will return to the study site on Day 7 to complete follow up assessments, on Day 28 for follow-up assessments including an X-Ray, and on Day 42 for the end-of-study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to sign the informed consent form (ICF) prior to study participation
* In the medical judgment of the Investigator, be a reasonably healthy adult 18 - 75 years of age, inclusive, and ASA Class I or II at the time of randomization
* Plan to undergo an elective primary unilateral, distal, first metatarsal bunionectomy with osteotomy and internal fixation under regional anesthesia, without collateral procedures or additional surgeries
* Have a BMI ≤ 39 kg/m2

Exclusion Criteria:

* Previous unilateral simple bunionectomy
* Has a planned concurrent surgical procedure that may impact pain scores, rescue medication use, or ability to fulfill the requirements of the protocol
* Concurrent painful condition
* Active skin disease or other clinically significant abnormality at the anticipated surgical site that could interfere with the planned surgery
* Known hypersensitivity or known allergy, as determined by the Investigator, to the ingredients (i.e., excipients) of the study drug or any peri- or postoperative medications used in this study
* History or clinical manifestation of significant medical, neuropsychiatric, or other condition that could preclude or impair study participation or interfere with study assessments
* History of malignant hyperthermia or glucose-6-phosphate dehydrogenase deficiency
* History or evidence of impaired liver function (e.g., ALT > 3 × upper limit of normal [ULN] or total bilirubin > 2 × ULN), active hepatic disease, or cirrhosis
* History or evidence of impaired renal function (e.g., creatinine > 1.5 × ULN)
* History of malignancy in the past year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized in situ carcinoma of the cervix
* Has or has had active COVID-19 infection within 3 months prior to surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
AUC72 | 72 hours post-operative
  Pain score through 72 hours post-operative

SECONDARY OUTCOMES:
Opioid use (MME) | 72 hours post-operative
  Opioid use through 72 hours post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, Study Chair — Cali Biosciences
Locations (3):
- United States (3):
  - Arizona Research Center, Phoenix, Arizona
  - Trovare Clinical Research, Bakersfield, California
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No